CLINICAL TRIAL: NCT04187443
Title: A Multicenter, Open-label, Dose Escalation Study Assessing the Safety and Treatment Effects of MS-553 in Diabetic Retinopathy Patients With Central Involved Macular Edema
Brief Title: MS-553 in Diabetic Retinopathy Patients With Central Involved Macular Edema
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen MingSight Relin Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Fountain Medical Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: MingSight Pharmaceuticals, Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001-CN
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Macular Edema; Macular Edema; Type 2 Diabetes With Diabetic Macular Edema; Type 1 Diabetes With Diabetic Macular Edema; Diabetic Retinopathy
Keywords: Diabetic Macular Edema; Macular Edema; Center-involved Diabetic Macular Edema; Center-involved DME; DME; Diabetic Retinopathy
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MS-553 low dose (Experimental): low dose of MS-553 taken orally
  Interventions: Drug: MS-553
- MS-553 mid dose (Experimental): mid dose of MS-553 taken orally
  Interventions: Drug: MS-553
- MS-553 high dose (Experimental): high dose of MS-553 taken orally
  Interventions: Drug: MS-553

INTERVENTIONS:
Drug: MS-553 — MS-553

SUMMARY:
This is an open label dose-escalation study to evaluate the safety and treatment benefits of MS-553 in treatment-naive diabetic retinopathy patients with central involved macular edema. Fifteen subjects with diabetic macular edema will be enrolled into each of three dose cohorts and will receive oral administration of MS-553 for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or type 2) according to ADA or WHO diabetic diagnosis criteria
* Subject has the ability to follow the study instructions and is likely to complete all required study procedures and visits;
* All males and females must consent to pregnancy prevention during the study and qualified measures of birth control. All females of childbearing potential must consent to a pregnancy test before entering the study.
* Presence of central involved macular edema associated with diabetic retinopathy, i.e. diabetic macular edema (DME), as assessed by spectral domain optical coherence tomography (sd-OCT) of the central retina subfield thickness (CRT) at the Screening Visit (Centration must be confirmed by Investigators with signatures);
* Best Corrected Visual Acuity (BCVA) score ≥ 34 letters (approximately 20/200 to 20/20 Snellen equivalent or better) using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity protocol, and assessed at the Screening Visit Visual acuity (VA);
* Confirmation by the investigator that laser photocoagulation and anti-VEGF treatments are either declined by the patients or not needed and can be withheld for at least 3 months after the Screening Visit;
* Ocular media and pupil dilation adequate to permit good quality retinal imaging as assessed at Screening Visit.

Exclusion Criteria:

* Subjects with unstable metabolic or blood pressure control
* Subject with emaciation or obesity at Screening Visit: body mass index (BMI) <18.5kg/m2 or >28kg/m2
* Current use or likely need for medications know to be toxic to the lens, retina or optic nerve, including Deferoxamine, Chloroquine / hydroxychloroquine (Plaquenil), Tamoxifen, Phenothiazines and Ethambutol -
* History of myocardial infarction or other cardiac event requiring hospitalization (unstable angina pectoris, etc.), cerebrovascular accident, transient ischemic attack, treatment for acute congestive heart failure or any arrhythmia within 4-months prior to Screening Visit;
* Any situation that may in the opinion of the investigator preclude the safe administration of the study medication, adherence to the scheduled study visits, safe participation in the study or affect the results of the study as assessed at Screening Visit;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | Baseline to Day 56

SECONDARY OUTCOMES:
Mean change in the central retina subfield thickness (CRT) | Baseline to Day 56
Mean change in the retinal volume | Baseline to Day 56
Proportion of patients with >20% reduction in CRT | Baseline to Day 56
Proportion of patients with resolution of central involved macular edema | Baseline to Day 56
Average mean change in best corrected visual acuity | Baseline to Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zhang, MD, Study Director — Shenzhen MingSight Relin Pharmaceuticals Co., Ltd.
Locations (3):
- China (3):
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Shanghai General Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No